CLINICAL TRIAL: NCT04205071
Title: Pilot Trial of Acute Effect of Lorcaserin to Reduce Patient-Reported Symptoms of Taxane- and Oxaliplatin-Induced Peripheral Neuropathy
Brief Title: Lorcaserin in Treating Chemotherapy-Induced Peripheral Neuropathy in Patients With Stage I-IV Gastrointestinal or Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decision
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Maryam Lustberg, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19085; NCI-2019-03368 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016058 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-12-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Chemotherapy-Induced Peripheral Neuropathy; Digestive System Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lorcaserin) (Experimental): Patients receive lorcaserin PO on day 1. The starting dose of lorcaserin will be 10 mg.
  Interventions: Drug: Lorcaserin; Drug: Lorcaserin Hydrochloride; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Lorcaserin — Given PO
Drug: Lorcaserin Hydrochloride — Given PO
  Other Names: LORCASERIN HYDROCHLORIDE ANHYDROUS
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies how well lorcaserin works in treating chemotherapy-induced peripheral neuropathy in patients with stage I-IV gastrointestinal or breast cancer. Chemotherapy-induced peripheral neuropathy is a nerve problem that causes pain, numbness, tingling, swelling, or muscle weakness in different parts of the body. This condition can occur in patients who have received taxane chemotherapy drugs, or the chemotherapy drug oxaliplatin. Lorcaserin may improve chemotherapy-induced peripheral neuropathy by reducing pain, preventing or relieving joint symptoms, and improving balance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate preliminary efficacy of lorcaserin to improve balance decrements in patients with chronic chemotherapy-induced peripheral neuropathy (CIPN).

SECONDARY OBJECTIVES:

I. To evaluate patient reported outcomes (PROs) after a one time dose of lorcaserin in patients with chronic CIPN.

OUTLINE:

Patients receive lorcaserin orally (PO) on day 1.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient with known diagnosis of gastrointestinal (GI) cancer or breast cancer stages I-IV
* Prior exposure to paclitaxel or oxaliplatin within last 24 months
* Have symptomatic CIPN confirmed by self-report, as demonstrated by PRO measure, CIPN-20
* If a female subject is with child bearing potential, she must have a negative pregnancy test at screening
* Female subjects of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 3 months after completion of study treatment administration. Adequate contraception includes methods such as oral contraceptives, double barrier method (condom plus spermicide or diaphragm), or abstaining from sexual intercourse
* Be willing and able to understand and sign the written informed consent document

Exclusion Criteria:

* Is beyond 24 months out from completion of oxaliplatin or paclitaxel
* Is asymptomatic for CIPN
* Is currently pregnant or breast feeding as there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lorcaserin
* Has any other medical or psychiatric condition that in the opinion of the investigator would make the study therapy unsafe for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the improvement in balance for patients with chronic CIPN | Up to 4 weeks
  Will be evaluated using a measure of postural control: root-mean-squared amplitude of center of pressure (COP) excursion for the medial-lateral axis of the body .

SECONDARY OUTCOMES:
Improvement in patient-reported chemotherapy-induced peripheral neuropathy symptoms | Baseline up to 4 weeks
  Evaluate using Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF is an additional PRO. It is a validated instrument that has been used to evaluate pain symptoms and functional capacity in our target population.45

OTHER OUTCOMES:
Nerve conduction test (NCT) result analysis | Baseline up to 4 weeks
  The study will compare baseline variables of patients with abnormal NCT results to those with normal NCT results. Will present descriptive statistics and perform t-tests comparing the two groups with respect to demographics (age, BMI), RMSml, and patient-reported outcomes (CIPN 20, BPI-SF).

CONTACTS AND LOCATIONS:
Overall Officials: Maryam B Lustberg, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu